CLINICAL TRIAL: NCT01684826
Title: Clinical Validation and Evaluation of ClarityIQ Cardiac Image Processing for Cardiac Angiography and Intervention
Brief Title: X-ray Dose Reduction Study for Cardiac Angiography and Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: XCY607-100084
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Vascular Diseases
Keywords: X-rays; Image processing; Cardiovascular procedure
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ClarityIQ (Experimental): Angiographic run with new algorithm and low dose (50% dose)
  Interventions: Radiation: Angiographic run with new algorithm and low dose (50% dose)
- AlluraXper (Experimental): Angiographic run with predecessor algorithm and dose (100% dose)
  Interventions: Radiation: Angiographic run with predecessor algorithm and dose (100%)

INTERVENTIONS:
Radiation: Angiographic run with new algorithm and low dose (50% dose) — Angiographic run with new algorithm and low dose (50% lower dose compared to Xper)
  Other Names: ClarityIQ
  Arms: ClarityIQ
Radiation: Angiographic run with predecessor algorithm and dose (100%) — Angiographic run with predecessor algorithm and dose (100% dose)
  Other Names: AlluraXper
  Arms: AlluraXper

SUMMARY:
ClarityIQ is a novel X-ray imaging technology, that combines advanced real-time image noise reduction algorithms, with state-of-the-art hardware to reduce patient entrance dose significantly. This is realized by anatomy-specific optimization of the full acquisition chain (grid switch, beam filtering, pulse width, spot size, detector and image processing engine) for every clinical task individually. Furthermore, smaller focal spot sizes and shorter pulses are used, which are known to positively influence image quality . The final effect on the clinical image quality is investigated in this study.

DETAILED DESCRIPTION:
Fluoroscopically guided procedures are associated with a risk of radiation injury to the skin, caused by high peak skin dose. The increasingly complex nature of many of the interventions performed requires the use of significant amounts of radiation for their completion. Of particular relevance to dose reduction concerns are obese patients, for whom additional radiation is often necessary to obtained sufficient diagnostic quality, as well as patients suffering from chronic total coronary occlusions (CTO), for whom long procedures with extended radiation time and contrast usage are common.

In order to introduce a dose reduction technology the most important aspect is to validate the diagnostic image information. Philips has developed a new algorithm that is capable to process images with similar image quality but acquired at lower dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age undergoing coronary angiography

Exclusion Criteria:

* Patients not willing or unable to give consent to participate
* Patients already involved in a clinical trial
* Patients under the age of 18
* Pregnant women and breastfeeding women
* Patients with severe kidney disease (eGFR < 60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry Suryapranata, Prof Dr., Principal Investigator — Radboud University Nijmegen Medical Center
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of patients occurred between 11 September and 23 November 2012.
Pre-assignment Details: 50 patients enrolled the study one subject withdrew consent.
Groups:
- AlluraXper-ClarityIQ: Angiogram with AlluraXper followed by angiogram with ClarityIQ
Period: Overall Study
Arm/Group | AlluraXper-ClarityIQ
Started | 49
Collected Dose and Image Information | 39
Completed | 39
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | AlluraXper-ClarityIQ
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 27
Region of Enrollment [Number; unit: participants]
  Netherlands | 49

OUTCOME MEASURES:

1. Primary Outcome: Image Quality
Description: Overall proportion where diagnostic image quality of ClarityIQ is scored equal or better compared to AlluraXper by the blinded readers. Reading is performed by simultaneous visual comparison of the image quality of AlluraXper and ClarityIQ by multiple blinded reviewers.The images are presented in a randomized order.
  The hypothesis is that the overall proportion where diagnostic image quality of ClarityIQ is scored equal or better is ≥ than 0.80. Combined for all raters, the lower bound of the one-sided 95% CI (lower bound of the two-sided 90% CI)is used.
Time Frame: 1 day
Population: All patient with recorded dose information and images for both angiograms were used.
Measure: Mean (90% Confidence Interval); unit: proportion of readers
Arm/Group | AlluraXper-ClarityIQ
Number analyzed (Participants) | 39
proportion of readers | 0.85 [0.82 to 0.89]

2. Secondary Outcome: Radiation Dose Measurements: Dose Area Product (DAP)
Description: Percentage of change of ClarityIQ vs. AlluraXper in Dose Area Product (DAP) calculated by DAP/frame. Negative percentage means a reduction in dose for ClarityIQ vs. AlluraXper.
Time Frame: Participants were followed for the duration of the procedure
Population: all patients with recorded dose information and images for both angiograms were included (n=39)
Measure: Mean (Standard Deviation); unit: percentage of dose change
Arm/Group | AlluraXper-ClarityIQ
Number analyzed (Participants) | 39
percentage of dose change | -52 (14)

3. Other Pre Specified Outcome: Radiation Dose Measurements: Air Kerma (AK)
Description: Percentage of change of ClarityIQ vs. AlluraXper in Air Kerma (AK) calculated by AK/frame. Negative percentage means a reduction in dose for ClarityIQ vs. AlluraXper.
Time Frame: Participants were followed for the duration of the procedure
Population: all patients with recorded dose information and images for both angiograms were included (n=39)
Measure: Mean (Standard Deviation); unit: percentage of dose change
Arm/Group | AlluraXper-ClarityIQ
Number analyzed (Participants) | 39
percentage of dose change | -53 (12)

ADVERSE EVENTS:
Time Frame: During procedure
Arm/Group | AlluraXper-ClarityIQ
Serious Adverse Events (participants affected / at risk) | 2/49
Other Adverse Events (participants affected / at risk) | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AlluraXper-ClarityIQ (N=49)
Ventricle Fibrillations (VF) (Cardiac disorders) | 1 (1) — defibrillation is done with 150 J
Type 2 Aorta dissection (Cardiac disorders) | 1 (1) — patient has atypical complaints. Suspected ACS. Troponin negative. Bloodpressure declines. Remaining contrast extra vasal (contrast injection in false lumen). Emergency CT scan made. Confirmed Aorta Dissection. Patient underwent emergency surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less